CLINICAL TRIAL: NCT06315894
Title: Design and Implementation of a Supervised Computerized Active Program (SuperCAP) for Improvement of Cognitive, Emotional, and Functional Status in People With Post-COVID Syndrome. SuperCAP Study
Brief Title: Supervised Computerized Active Program for People With Post-COVID Syndrome (SuperCAP Study)
Acronym: SuperCAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Collaborators: Institut de Recerca de la SIDA IrsiCaixa (Unknown); Germans Trias i Pujol Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI-22-191
Record Dates: First submitted 2024-03-15; First posted 2024-03-18 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Post-COVID Condition
Keywords: Long COVID (LC); Post-Acute COVID-19 Syndrome (PACS); Post-Acute Sequelae of COVID-19 (PASC); Post-Acute Sequelae of SARS-CoV-2 (PASS); Post-COVID Condition (PCC); Post-COVID Syndrome (PCS)
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): People with post-COVID syndrome following the intervention
  Interventions: Device: SuperCAP Program
- Control (No Intervention): People with post-COVID syndrome not following the intervention

INTERVENTIONS:
Device: SuperCAP Program — Distance program including tasks and exercises to improve cognitive, emotional, and functional status.
  The intervention will be applied via cell phone and will have a duration of 3 months (12 weeks).
  Tasks and exercises will be performed 5 days per week. Contents of the program will include daily exercises, daily games, daily videos, and weekly videos.
  They will address cognitive functions, daily habits, and lifestyle factors in general.
  Compliance will be monitored to control the adherence to the intervention. The program has been designed specifically for people with post-COVID syndrome.
  Arms: Experimental

SUMMARY:
SuperCAP study is a project aimed at designing and implementing an online program for improvement of cognitive, emotional, and functional status in post-COVID condition.

DETAILED DESCRIPTION:
SuperCAP study will include 2 stages.

Stage 1 will involve the composition of a focus group previous to the effectiveness study development.

The work with this focus group will have several aims, among them, mainly, to participate in the design of the intervention program, and to provide feedback on the study follow-up.

Stage 2 will include the effectiveness study. This stage will comprise the initiation of the intervention program, study follow-up, and dissemination of the results in the end of the project.

Two study groups will participate: the Intervention Group and the Control Group.

The Intervention Group will be comprised by people with post-COVID condition who will follow the intervention program proposed.

The Control Group will be comprised by people with post-COVID condition who will not follow the program.

Both groups will fulfill the same study participation criteria.

The intervention will consist of the follow-up of a distance program via mobile/tablet. This program will integrate different games and exercises always with the objective of stimulating the cognitive functioning and the emotional status.

ELIGIBILITY:
Inclusion Criteria:

* Presenting Post-COVID Syndrome, defined as presenting 3 or more symptoms associated with post-COVID condition for at least 3 months.
* Age of 18-65 years old.
* Presence of self-reported cognitive complaints associated with post-COVID infection.
* Positive and favorable attitude on the use of electronic devices.
* Will to participate in a stimulation program for improvement of cognitive symptoms.
* Availability of cell phone and computer or tablet with the minimum technical features considered.

Exclusion Criteria:

* Inability to undergo the neuropsychological tests or complementary study assessments.
* Current participation in a trial or program for improvement of post-COVID symptoms.
* Any condition that in the opinion of the investigator would make study participation unsafe, complicate interpretation of study outcome data, interfere with achieving the study objectives, or otherwise could impair the subject's ability to complete the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
Change in Self-reported Cognitive Functioning | From Baseline to Week 12
  Understanding and Communicating Scale (D1) from WHODAS 2.0 questionnaire. Scores from 0 to 20. Lower scores indicate better functioning, higher scores worse functioning.

SECONDARY OUTCOMES:
Change in Performance-based Cognitive Functioning | From Baseline to Week 12
  NPZ12, global neuropsychological measure. Scores from -5 to +5. Lower scores indicate worse functioning, higher scores better functioning.
Change in Depression Symptoms | From Baseline to Week 12
  PHQ-9 questionnaire. Scores from 0 to 27. Lower scores indicate fewer symptoms, higher scores more symptoms.
Change in Anxiety Symptoms | From Baseline to Week 12
  GAD-7 questionnaire. Scores from 0 to 21. Lower scores indicate fewer symptoms, higher scores more symptoms.
Change in Daily Activities Functioning | From Baseline to Week 12
  IADL scale. Scores from 0 to 20. Lower scores indicate better functioning, higher scores worse functioning.
Change in Physical Activity | From Baseline to Week 12
  IPAQ questionnaire. Scores from 0 to undetermined (total days, hours, minutes reported). Lower scores indicate worse activity, higher scores better activity.
Change in Quality of Life | From Baseline to Week 12
  EuroQoL-5D scale. Scores from 0 to 100. Lower scores indicate worse quality of life, higher scores better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Germans Trias I Pujol Hospital, Badalona, Barcelona, Spain